CLINICAL TRIAL: NCT04253418
Title: Prospective, Open Label, Multi-Center, Non-Significant Risk Study of Nano-Pulse Stimulation™ (NPS™ ) Technology in Healthy Adults With Sebaceous Hyperplasia
Brief Title: Nano-Pulse Stimulation (NPS) in Sebaceous Hyperplasia Optimization Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study enrollment was halted due to a business decision by the Sponsor to focus resources on other clinical areas outside of dermatology.
Sponsor: Pulse Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP-SH-009
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Sebaceous Hyperplasia; Skin Abnormalities; Skin Lesion
MeSH Terms: conditions — Skin Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Nano-Pulse Stimulation (NPS) Treated Lesion (Experimental): Nano-Pulse Stimulation of target lesion.
  Interventions: Device: Nano-Pulse Stimulation (NPS)

INTERVENTIONS:
Device: Nano-Pulse Stimulation (NPS) — Electrical pulses (nanosecond duration) applied directly to target SH lesions using sterile single-patient use treatment tips with microneedles.

SUMMARY:
Primary study objective is to evaluate the optimization of Nano-Pulse Stimulation (NPS) energy settings for lesion clearance of Sebaceous Hyperplasia (SH) lesions from facial areas of healthy adult subjects.

DETAILED DESCRIPTION:
* Evaluate lesion clearance of treated facial Sebaceous Hyperplasia lesions using multiple sized treatment tips with microneedles.
* Evaluate lesion clearance of the treated Sebaceous Hyperplasia lesions using multiple energy settings levels at various time points.
* Evaluate skin effects and adverse event rate.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female between 18 and 75 years of age
* Voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.
* Understanding of the clinical investigation, agree to cooperate with the investigational procedures and are willing to return for all the required follow-up visits.
* Understands that SHs are to be treated in a single treatment session is aware that they may receive a second treatment at their third study visit
* Must be able to visit clinic site at 7-, 30-, 60-days post-primary treatment of SH lesion and at 30- and 60-days post-retreatment.
* Clinically diagnosis of typical sebaceous hyperplasia.
* Minimum of four SH lesions.
* Undergo all study procedures including consent for photographs of the treated SH sites.
* Agrees to refrain from using all other SH lesion removal products or treatments (topical medication including over-the-counter medications) during the study period.

Exclusion Criteria:

* Implantable electronic devices (i.e., pacemaker, implantable cardioverter defibrillator)
* Active infection or history of infection in designated test area within 90 days prior to first treatment.
* Not willing or able to sign the Informed Consent.
* Known to be immune-compromised.
* Known to be a keloid producer.
* Taking blood thinning medications.
* Insulin dependent, Type I diabetics.
* Allergies to Lidocaine or Lidocaine-like products.
* Employed by the sponsor, clinic site, or entity associated with the conduct of the study.
* Have any condition or situation which, in the Investigator's opinion, puts the subject at significant risk, could confound the study results, or may interfere significantly with the subject's participation in the study.
* Known prior inability to complete required study visits during treatment period.
* Use of any other investigational drug, therapy, or device within the past 30 days of enrollment or concurrent participation in another research study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
SH Lesion Clearance Rate | 60-days post-last NPS treatment
  Clearance of SH lesions treated with NPS as rated by investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Nuccitelli, PhD, Study Chair — Pulse Biosciences, Inc.
Locations (6):
- United States (6):
  - Clear Dermatology & Aesthetics Center / InvestigateMD, Scottsdale, Arizona
  - Laser and Skin Surgery Center of Northern California, Sacramento, California
  - AVA MD, Santa Monica, California
  - Capital Laser & Skin Care, Chevy Chase, Maryland
  - United Skin Physicians, Chestnut Hill, Massachusetts
  - Dermatology, Laser & Vein Specialists of the Carolinas, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No